CLINICAL TRIAL: NCT02831101
Title: Impact of Sufentanil on the Depth of Sedation Measured by Bispectral Index During Induction of Anaesthesia With Propofol in the Elderly - a Randomised Trial
Brief Title: Sufentanil Bispectral Index Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christopher Lysakowski, MD PD, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: CER 11-25, NAC 11-78
Record Dates: First submitted 2016-07-01; First posted 2016-07-13 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Loss of Consciousness
Keywords: BIS; Elderly; Propofol; Sufentanil; Loss of consciousness
MeSH Terms: conditions — Unconsciousness | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sufentanil (Experimental): Sufentanil intravenously, continuously with effect-site concentration of 0.3 ng/ml until the end of the study
  Interventions: Drug: Sufentanil
- Placebo (Other): Saline intravenously, continuously with the same effect-site concentration as sufentanil (recorded on administration device) until the end of the study
  Interventions: Drug: Placebo
- Propofol (No Intervention): Open administration using a separate target controlled infusion system and the PK/PD model by Schnider. Initial effect-site concentration 0.5 mcg/ml increased by 0.5 mcg/ml until LOC

INTERVENTIONS:
Drug: Sufentanil — To evaluate, in the elderly, the impact of a concomitant administration of sufentanil during a step-wise propofol induction of anaesthesia on the depth of sedation measured using BIS and clinical sedation score.
  Arms: Sufentanil
Drug: Placebo — To evaluate presence or absence of strong opioid (sufentanil) on BIS values in the elderly during propofol induction until the loss of consciousness
  Arms: Placebo

SUMMARY:
We compared BIS values during propofol stepwise induction with or without concomitant sufentanil in patients ≥ 65 years .

DETAILED DESCRIPTION:
Bispectral index (BIS) is widely used to estimate the depth of anesthesia. In clinical studies, a large variability of BIS has been observed. Several factors may be responsible for this inconsistency. We were able to show that in elderly patients (average age 78 years) receiving increasing doses of propofol alone a BIS values at loss of consciousness (LOC) were about 30% higher compared with young patients (average age 35 years). We showed also that in young patients (average age 48 years) the BIS values at LOC were significantly higher in those receiving sufentanil concomitantly with propofol compared with those who had received propofol alone. It remains unknown, however, whether these data from young surgical patients are applicable to a population of elderly patients. It may be argued that in the elderly receiving propofol, the impact of advance age was so important that any addition of an opioid would not further disturb the sedation-monitor balance. Alternatively, it may be expected that in the elderly receiving an opioid added to propofol the impact of both drugs on sedation will be additive and that previous observations from younger patients will be further exaggerated. The impact of advance age and presence or absence of sufentanil during propofol induction on BIS values at LOC was investigated in this trial.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥65 years

Exclusion Criteria:

* History of heart disease
* History of renal disease
* History of psychiatric
* Obesity
* Allergy to propofol or sufentanil

Ages: 70 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
BIS at baseline | BIS values at baseline before administration of any study drugs
  BIS values in awake patient in supine position, eyes closed, quiet environment
BIS and sufentanil | BIS values 10 min after steady state concentration of sufentanil
  BIS values recorded after the steady state concentration was obtained and kept during 10min.
BIS and propofol | BIS values after steady state concentration of propofol
  Propofol was administrated step-wise by increasing concentration of 0.5mcg/ml (0.5, 1.0, 1.5 etc.). After each steady state that was kept during 5 min, BIS values were recorded
BIS and LOC | BIS values at loss of consciousness
  BIS values were recorded at LOC, that was estimated using a OAA/S scale, a 0-5 point scale, 5 corresponds to a fully awake state, a score of 0 to a completely unresponsive state. A score <2 (absence of response to mild prodding or shaking was regarded as LOC. Blinded to study drug investigator evaluated all sedation scores.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Valence T, Elia N, Czarnetzki C, Dumont L, Tramer MR, Lysakowski C. Effect of sufentanil on bispectral index in the elderly. Anaesthesia. 2018 Feb;73(2):216-222. doi: 10.1111/anae.14102. Epub 2017 Nov 3. PMID 29098683